CLINICAL TRIAL: NCT01985867
Title: Effectiveness of Lactobacillus Casei Rhamnosus Lcr35 in the Management of Children With Functional Constipation: a Randomized, Double-blind, Placebo- Controlled Trial.
Brief Title: Lcr35 for Children With Functional Constipation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, Katarzyna Wojtyniak, MD, Medical University of Warsaw
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1-2013
Record Dates: First submitted 2013-10-30; First posted 2013-11-15 (Estimated); Results first posted 2023-05-17 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-05

CONDITIONS: Constipation
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lactobacillus casei rhamnosus Lcr35 (Experimental): Eligible children will receive Lactobacillus casei rhamnosus Lcr35 8×10^8 colony forming units (CFU), twice daily, orally for 4 weeks
  Interventions: Dietary Supplement: Lactobacillus casei rhamnosus Lcr35
- Placebo (Placebo Comparator): Eligible children will receive placebo (maltodextrin), twice daily, orally for 4 weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Lactobacillus casei rhamnosus Lcr35 — Eligible children will receive Lactobacillus casei rhamnosus Lcr35 (8×10^8 CFU, twice daily, orally for 4 weeks)
  Arms: Lactobacillus casei rhamnosus Lcr35
Dietary Supplement: Placebo — Eligible children will receive placebo (maltodextrin), twice daily, orally for 4 weeks
  Arms: Placebo

SUMMARY:
The aim of this study is to assess the effectiveness of Lactobacillus casei rhamnosus Lcr35 administration for the treatment of functional constipation in children.

DETAILED DESCRIPTION:
Functional constipation is a common problem which affects over 3% of children. The standard treatment does not provide sustained relief of symptoms. As a consequence, there is interest in other therapeutic options. Previously, one small (n=40) randomized controlled trial (RCT) involving 27 children showed that Lactobacillus rhamnosus casei Lcr35 compared with placebo increased treatment success defined as ≥ 3 spontaneous defecations per week with no episodes of faecal soiling, increased the defecation frequency, reduced the frequency of abdominal pain, reduced the use of glycerin enemas during the four weeks of therapy, and decreased the percentage of hard stools. However, there was no difference between groups in the use of lactulose or the number of episodes of faecal soiling. Available evidence is insufficient to draw meaningful conclusion. Further studies are needed.

ELIGIBILITY:
Inclusion Criteria:

* Children below 5 years of age
* Functional constipation according to Rome III criteria i.e. 1 month of at least 2 of the following:

  * Two or fewer defecations per week
  * At least 1 episode per week of incontinence after the acquisition of toileting skills
  * History of excessive stool retention
  * History of painful or hard bowel movements
  * Presence of a large fecal mass in the rectum
  * History of large- diameter stools that may obstruct the toilet

Exclusion Criteria:

* Irritable bowel syndrome
* Mental retardation
* Endocrine disease (e.g. hypothyroidism)
* Organic cause of constipation (e.g. Hirschsprung disease)
* Spinal anomalies
* Anatomic defects of the anorectum
* History of previous gastrointestinal surgery
* Functional nonretentive fecal incontinence
* Use of drugs that influence gastrointestinal motility

Max Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 94 (Actual)
Dates: Start 2013-11; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hania Szajewska, MD, Principal Investigator — Medical University of Warsaw
Locations (1):
- Department of Pediatrics, Medical University of Warsaw, Warsaw, Poland

REFERENCES:
- [Derived] Wojtyniak K, Horvath A, Dziechciarz P, Szajewska H. Lactobacillus casei rhamnosus Lcr35 in the Management of Functional Constipation in Children: A Randomized Trial. J Pediatr. 2017 May;184:101-105.e1. doi: 10.1016/j.jpeds.2017.01.068. Epub 2017 Mar 8. PMID 28284477

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lactobacillus Casei Rhamnosus Lcr35 | Placebo
Started | 48 | 46
Completed | 41 | 40
Not Completed | 7 | 6
Not completed — Lost to Follow-up | 3 | 4
Not completed — Adverse Event | 3 | 2
Not completed — Lack of Efficacy | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lactobacillus Casei Rhamnosus Lcr35 | Placebo | Total
Number analyzed (Participants) | 48 | 46 | 94
Age, Continuous [Mean (Standard Deviation); unit: month] | 38.7 (12.1) | 37.3 (14.2) | 38 (13.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 26 | 52
  Male | 22 | 20 | 42
Region of Enrollment [Count of Participants; unit: Participants]
  Poland | 48 | 46 | 94
Age of onset of constipation [Mean (Standard Deviation); unit: months] | 24.0 (12.1) | 23.5 (12.9) | 23.77 (12.45)
Duration of constipation [Mean (Standard Deviation); unit: months] | 14.7 (9.1) | 13.8 (11.1) | 14.3 (10.1)
Stools per week [Mean (Standard Deviation); unit: Stools per week] | 1.6 (0.5) | 1.6 (0.5) | 1.6 (0.5)
Stool consistency, Bristol scale [Mean (Standard Deviation); unit: units on a scale] — The 7-point Bristol Stool Form Scale (BSFS), which refers to 7 pictures of different forms of stool, is a commonly used instrument to assess stool consistency.
  Bristol Stool Form Scale:
  Type 1- Separate hard lumps, like nute (hard to pass); Type 2- Sausage- shaped but lumpy; Type 3- Like a sausage but with cracks on the surface; Type 4- Like a sausage or snake, smooth and soft; Type 5- Soft blobs with clear-cut edges; Type 6- Fluffy pieces with ragged edges, a mushy stool; Type 7- Watery, no solid pieces. Entirely Liquid.
  units on a scale | 1.5 (1.0) | 1.7 (0.9) | 1.6 (0.9)
Fecal soiling [Count of Participants; unit: Participants] | 21 | 21 | 42
Pain during defecation [Count of Participants; unit: Participants] | 47 | 44 | 91
Withholding behavior [Count of Participants; unit: Participants] — Parents assess witholding behaviour like rock back and forth while stiffening buttocks and legs, arch back, cross legs, stand on tiptoes, and wriggle or fidget, or squat or get into other unusual positions.
  Participants | 44 | 41 | 85
Abdominal pain [Count of Participants; unit: Participants] | 27 | 29 | 56
Blood in the stool [Count of Participants; unit: Participants] | 17 | 14 | 31
Previous treatment for intestinal constipation [Count of Participants; unit: Participants] | 40 | 37 | 77
Rectal impaction [Count of Participants; unit: Participants] | 35 | 35 | 70

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Success (≥3 Spontaneous Defecations Per Week With no Fecal Soiling
Time Frame: in the fourth week of the intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Lactobacillus Casei Rhamnosus Lcr35 | Placebo
Number analyzed (Participants) | 48 | 46
Participants | 24 | 28
Statistical Analysis 1: Comparison: Lactobacillus Casei Rhamnosus Lcr35 vs Placebo; Test type: Superiority or Other; p = 0.399, risk analysis (prospective); Risk Ratio (RR) = 1.19, 95% CI 2-sided [0.24 to 1.5]

2. Secondary Outcome: Stool Consistency at Week 4
Description: Stool consistency scores were determined using the 7-point Bristol Stool Form Scale (1 for hard lumps to 7 for watery stools).
  For single value median was calculated.
Time Frame: during fourth week of intervention
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Lactobacillus Casei Rhamnosus Lcr35 | Placebo
Number analyzed (Participants) | 41 | 40
units on a scale | 3.5 [2.8 to 4.0] | 3.7 [3.0 to 4.0]
Statistical Analysis 1: Comparison: Lactobacillus Casei Rhamnosus Lcr35 vs Placebo; Test type: Superiority or Other; p = 0.589, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 0.2, 95% CI 2-sided [-0.6 to 0.7]

3. Secondary Outcome: Defecation Frequency at Week 4
Description: For single value median was calculated.
Time Frame: during fourth week of intervention
Measure: Median (Inter-Quartile Range); unit: defecations per week
Arm/Group | Lactobacillus Casei Rhamnosus Lcr35 | Placebo
Number analyzed (Participants) | 41 | 40
defecations per week | 4.0 [3.0 to 5.0] | 6.0 [4.0 to 9.0]
Statistical Analysis 1: Comparison: Lactobacillus Casei Rhamnosus Lcr35 vs Placebo; Test type: Superiority or Other; p = 0.005, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 2.0, 95% CI 2-sided [0.5 to 4.0]

4. Secondary Outcome: Fecal Soiling Episodes at Week 4
Description: For single value median was calculated.
Time Frame: during fourth week of intervention
Measure: Median (Inter-Quartile Range); unit: fecal soiling episodes
Arm/Group | Lactobacillus Casei Rhamnosus Lcr35 | Placebo
Number analyzed (Participants) | 41 | 40
fecal soiling episodes | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0]
Statistical Analysis 1: Comparison: Lactobacillus Casei Rhamnosus Lcr35 vs Placebo; Test type: Superiority or Other; p = 0.659, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 0.0, 95% CI 2-sided [0.0 to 0.0]

5. Secondary Outcome: Number of Defecations That Were Painful at Week 4
Description: Pain reported by child or symptoms of pain observed by parents. For single value median was calculated.
Time Frame: during fourth weeks of intervention
Measure: Median (Inter-Quartile Range); unit: painful defecations
Arm/Group | Lactobacillus Casei Rhamnosus Lcr35 | Placebo
Number analyzed (Participants) | 41 | 40
painful defecations | 0.0 [0.0 to 1.0] | 0.0 [0.0 to 1.0]
Statistical Analysis 1: Comparison: Lactobacillus Casei Rhamnosus Lcr35 vs Placebo; Test type: Superiority or Other; p = 0.790, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 0.0, 95% CI 2-sided [0.0 to 0.0]

6. Secondary Outcome: Abdominal Pain at Week 4
Description: Abdominal pain reported by child or symptoms of pain observed by parents. For single value median was calculated.
Time Frame: during fourth weeks of intervention
Measure: Median (Inter-Quartile Range); unit: abdominal pain episodes
Arm/Group | Lactobacillus Casei Rhamnosus Lcr35 | Placebo
Number analyzed (Participants) | 41 | 40
abdominal pain episodes | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0]
Statistical Analysis 1: Comparison: Lactobacillus Casei Rhamnosus Lcr35 vs Placebo; Test type: Superiority or Other; p = 0.698, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 0.0, 95% CI 2-sided [0.0 to 0.0]

7. Secondary Outcome: Number of Participants With Use of Laxatives
Time Frame: during 4 weeks of intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Lactobacillus Casei Rhamnosus Lcr35 | Placebo
Number analyzed (Participants) | 41 | 40
Participants | 18 | 10
Statistical Analysis 1: Comparison: Lactobacillus Casei Rhamnosus Lcr35 vs Placebo; Test type: Superiority or Other; p = 0.120, risk analysis (prospective); Risk Ratio (RR) = 2.3, 95% CI 2-sided [0.9 to 6.2]

8. Secondary Outcome: Number of Participants With Adverse Effects
Time Frame: during 4 weeks of intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Lactobacillus Casei Rhamnosus Lcr35 | Placebo
Number analyzed (Participants) | 41 | 40
Participants | 0 | 3
Statistical Analysis 1: Comparison: Lactobacillus Casei Rhamnosus Lcr35 vs Placebo; Test type: Superiority or Other; p = 0.116, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: Stool Consistency at Week 1
Description: as for outcome 2
Time Frame: during first week of intervention
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Lactobacillus Casei Rhamnosus Lcr35 | Placebo
Number analyzed (Participants) | 41 | 40
units on a scale | 3.6 [3.0 to 4.0] | 3.9 [2.8 to 4.3]
Statistical Analysis 1: Comparison: Lactobacillus Casei Rhamnosus Lcr35 vs Placebo; Test type: Superiority or Other; p = 0.612, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 0.5, 95% CI 2-sided [-0.6 to 0.8]

10. Secondary Outcome: Defecation Frequency at Week 1
Time Frame: during first week of intervention
Measure: Median (Inter-Quartile Range); unit: defecations per week
Arm/Group | Lactobacillus Casei Rhamnosus Lcr35 | Placebo
Number analyzed (Participants) | 41 | 40
defecations per week | 5.0 [3.0 to 6.0] | 6.0 [5.0 to 8.2]
Statistical Analysis 1: Comparison: Lactobacillus Casei Rhamnosus Lcr35 vs Placebo; Test type: Superiority or Other; p = 0.004, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 1.0, 95% CI 2-sided [0.0 to 2.0]

11. Secondary Outcome: Fecal Soiling Episodes at Week 1
Time Frame: during first week of intervention
Measure: Median (Inter-Quartile Range); unit: fecal soiling episodes
Arm/Group | Lactobacillus Casei Rhamnosus Lcr35 | Placebo
Number analyzed (Participants) | 41 | 40
fecal soiling episodes | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0]
Statistical Analysis 1: Comparison: Lactobacillus Casei Rhamnosus Lcr35 vs Placebo; Test type: Superiority or Other; p = 0.708, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 0.0, 95% CI 2-sided [0.0 to 0.0]

12. Secondary Outcome: Pain During Defecation at Week 1
Description: Pain reported by child or symptoms of pain observed by parents. For single value median was calculated.
Time Frame: during first weeks of intervention
Measure: Median (Inter-Quartile Range); unit: painful defecations
Arm/Group | Lactobacillus Casei Rhamnosus Lcr35 | Placebo
Number analyzed (Participants) | 41 | 40
painful defecations | 0.0 [0.0 to 1.0] | 0.0 [0.0 to 2.0]
Statistical Analysis 1: Comparison: Lactobacillus Casei Rhamnosus Lcr35 vs Placebo; Test type: Superiority or Other; p = 0.522, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 0.0, 95% CI 2-sided [-1.0 to 1.0]

13. Secondary Outcome: Abdominal Pain at Week 1
Description: Abdominal pain reported by child or symptoms of pain observed by parents. For single value median was calculated.
Time Frame: during first weeks of intervention
Measure: Median (Inter-Quartile Range); unit: abdominal pain episodes
Arm/Group | Lactobacillus Casei Rhamnosus Lcr35 | Placebo
Number analyzed (Participants) | 41 | 4
abdominal pain episodes | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 1.0]
Statistical Analysis 1: Comparison: Lactobacillus Casei Rhamnosus Lcr35 vs Placebo; Test type: Superiority or Other; p = 0.185, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 0.0, 95% CI 2-sided [0.0 to 1.0]

14. Secondary Outcome: Flatulence at Week 4
Description: Flatulence reported by child or symptoms of pain observed by parents. For single value median was calculated.
Time Frame: during fourth weeks of intervention
Measure: Median (Inter-Quartile Range); unit: episodes of flatulence
Arm/Group | Lactobacillus Casei Rhamnosus Lcr35 | Placebo
Number analyzed (Participants) | 41 | 40
episodes of flatulence | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0]
Statistical Analysis 1: Comparison: Lactobacillus Casei Rhamnosus Lcr35 vs Placebo; Test type: Superiority or Other; p = 0.973, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 0.0, 95% CI 2-sided [0.0 to 0.0]

15. Secondary Outcome: Flatulence at Week 1
Description: Flatulence reported by child or symptoms of pain observed by parents. For single value median was calculated.
Time Frame: during first weeks of intervention
Measure: Median (Inter-Quartile Range); unit: episodes of flatulence
Arm/Group | Lactobacillus Casei Rhamnosus Lcr35 | Placebo
Number analyzed (Participants) | 41 | 40
episodes of flatulence | 0.0 [0.0 to 1.0] | 0.0 [0.0 to 0.2]
Statistical Analysis 1: Comparison: Lactobacillus Casei Rhamnosus Lcr35 vs Placebo; Test type: Superiority or Other; p = 0.642, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 0.0, 95% CI 2-sided [0.0 to 0.0]

ADVERSE EVENTS:
Time Frame: during 4 weeks of the intervention
Arm/Group | Lactobacillus Casei Rhamnosus Lcr35 | Placebo
Serious Adverse Events (participants affected / at risk) | 0/48 | 0/46
Other Adverse Events (participants affected / at risk) | 0/48 | 3/46
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lactobacillus Casei Rhamnosus Lcr35 (N=48) | Placebo (N=46)
change in the stool smell (Gastrointestinal disorders) | 0 (0) | 1 (1)
abdominal pain and flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1)
loss of appetite (Gastrointestinal disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Children were recruited in an academic center specialized in the management of children with constipation. Outcomes were evaluated only based on non-validated stool diaries completed by caregivers, except for stool consistency.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No